CLINICAL TRIAL: NCT07125300
Title: Efficacy of an Artificial Intelligence System for Lesion Detection and Characterization (CADe and CADx) During Colorectal Cancer Screening Colonoscopies: A Randomized Clinical Trial
Brief Title: A Study Comparing Standard and AI-Assisted Colonoscopies for Detecting and Characterizing Colorectal Lesions in Adults Aged 50-74 Undergoing Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Javier Santos Fernández (Other)
Responsible Party: Sponsor-Investigator, Javier Santos Fernández, Clinical Trials Coordinator, University Care Complex of Palencia
Organization: University Care Complex of Palencia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2024/023
Record Dates: First submitted 2025-07-25; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Neoplasms; Colorectal Cancer; Adenoma Colon Polyp
Keywords: Colorectal cancer screening; Colonoscopy; Artificial Intelligence; CADe; CADx
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional colonoscopy without AI assistance (No Intervention)
- AI-assisted colonoscopy (Experimental)
  Interventions: Diagnostic Test: Artificial Intelligence-Assisted Colonoscopy

INTERVENTIONS:
Diagnostic Test: Artificial Intelligence-Assisted Colonoscopy — The intervention involves the use of an artificial intelligence tool during screening colonoscopy. This system includes two integrated functions:
  * CADe (Computer-Aided Detection): Highlights suspected lesions in real time on the endoscopic video to assist in identifying polyps.
  * CADx (Computer-Aided Diagnosis): Provides real-time optical histology predictions to help distinguish between hyperplastic and adenomatous polyps.
  The AI system operates autonomously during the procedure and displays visual cues on the monitor to support the endoscopist in detecting and characterizing colorectal lesions.
  Arms: AI-assisted colonoscopy

SUMMARY:
The goal of this clinical trial is to determine whether using artificial intelligence (AI) can improve the detection and characterization of abnormal growths (polyps) during colonoscopy in adults aged 50 to 74 years who are undergoing colorectal cancer screening after a positive stool test.

The main questions it aims to answer are:

* Does AI assistance increase the detection of adenomas or advanced colorectal neoplasia?
* Does AI provide more accurate optical diagnosis of polyps compared to standard assessment by endoscopists?

Researchers will compare colonoscopies performed with AI assistance (using the CAD EYE™ system) to standard colonoscopies without AI to see if AI improves detection rates or diagnostic accuracy.

Participants will:

* Undergo a screening colonoscopy after a positive fecal immunochemical test (FIT)
* Be randomly assigned to either an AI-assisted or standard colonoscopy group
* Have any detected polyps removed and analyzed
* Receive either AI-based or physician-based optical diagnosis of polyps during the procedure

This study helps evaluate whether AI can make colonoscopies more effective and reduce unnecessary polyp removals.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 50 to 74 years
* Positive fecal immunochemical test (FIT) result (≥100 ng/mL)
* Scheduled for screening colonoscopy within a population-based colorectal cancer screening program
* Able and willing to provide written informed consent

Exclusion Criteria:

* Incomplete colonoscopy (e.g., failure to reach the cecum)
* Inadequate bowel preparation
* History of colorectal surgery
* Inability to provide informed consent

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
To compare the adenoma detection rate (ADR) and advanced colorectal neoplasia detection rate between conventional colonoscopy and AI-assisted colonoscopy. | During the screening colonoscopy visit (single time point assessment on the day of the procedure).

SECONDARY OUTCOMES:
To compare mean number of lesions between conventional colonoscopy and AI-assisted colonoscopy. | During the screening colonoscopy visit (single time point assessment on the day of the procedure).

CONTACTS AND LOCATIONS:
Locations (1):
- University Care Complex of Palencia, Palencia, Spain

IPD SHARING:
Plan to Share IPD: No